CLINICAL TRIAL: NCT06189196
Title: Effects of Blow Bottle Verses ACBTs Technique in Patients of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Maryam Riphah
Record Dates: First submitted 2023-08-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: COPD
Keywords: Active cycle of breathing technique; Breathlessness; Cough; Chronic Obstructive Pulmonary Disease,; Sputum; Quality Of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): BLOW BOTTLE
  Interventions: Device: BLOW BOTTLE
- Group B (Experimental): ACBT
  Interventions: Other: ACBT

INTERVENTIONS:
Device: BLOW BOTTLE — Blow Bottle PEP' is the cost-effective device comparative to other PEP devices. Treatment (CPT) along with BBPEP twice a day. Therapist made a cost-effective BBPEP which generates 10 cm of H2O PEP and it was given for 10 breaths, 3 sets with 5 second hold.
  Arms: Group A
Other: ACBT — Active cycle of breathing technique (ACBT) is an alternative airway clearance technique. A typical ACBT cycle consists of breathing control, three to four thoracic expansion exercises, and a forced expiratory technique (huffing). ACBT has been shown to improve short-term secretion clearance in patients with chronic lung disease. It is also flexible, tolerated, and accepted well by patients. Although ACBT is widely used in patients with respiratory conditions characterized by chronic sputum production.
  Arms: Group B

SUMMARY:
Chronic obstructive pulmonary disease is a common disease worldwide. Pulmonary rehabilitation is an important part to decrease the complications of COPD. Blow bottle technique is an economical and subjective technique promote the lung expansion, as compare to ACBTs. It used to treat the different complications in COPD patients and also decrease the dependency of patient. To find the comparative effects of blow bottle and active cycle of breathing on sputum diary, oxygen saturation, pulmonary function and quality of life among the patients of chronic bronchitis.

A randomized clinical trial will be conducted at Gulab Devi hospital Lahore. Through convenient sampling technique on 56 patients, allocated through simple random sampling through computer generated technique into group A and Group B. Group A will be treated with blow bottle technique and group B will be treated by with ACBTs. Pretreatment values will be recorded for BCSS for sputum, pulse oximeter, pulmonary function test and st. George for quality of life will be assessed before and after 8 weeks of the treatment. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be use within a group or between two groups.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is defined as chronic airflow obstruction that is progressive. Patients with chronic obstructive pulmonary disease (COPD) are highly susceptible from respiratory exacerbations from viral respiratory tract infections. The pathological consequences of the COPD inflammation Induce series of physiological changes which eventually impact the quality of life and survival in the natural progress of COPD. Elastin proteolysis results in reduction in elastic recoil Pressures in the lungs, also the integrity and movement Of air in the bronchioles results in significant airway narrowing with air-trapping in lungs.

COPD is an increasingly important cause of morbidity, disability, and mortality worldwide. Researcher aimed to estimate global, regional, and national COPD prevalence and risk factors to guide policy and population interventions. Chronic Obstructive Pulmonary Disease (COPD) is attributable to household air pollution and is known to increase the Disability Adjusted Life Years (DALYs), morbidity and mortality and women are most susceptible groups for the exposure. In order to understand the global risk among women with COPD due to exposure of household air pollutants.

Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality worldwide. Smoking remains the most important risk factor, but occupational exposures may play an essential role as well n 2019, Thirty-two sources of COPD prevalence rates, representing 17 countries and eight World Health Organization-classified regions, were identified and reviewed. Reported prevalence ranged from 0.23 to 18.3%. The lowest prevalence rates 0.2 to 2.5% were based on expert opinion. Sixteen studies had measured rates that could reasonably be extrapolated to an entire region or country.

The physiotherapist has a major role to assume in pre and post-exacerbation management of people with COPD and assess the patient and to put into place an individualized pulmonary rehabilitation program. In patients with a range of respiratory disorders such as chronic bronchitis, different technique are available for pulmonary rehabilitation, such as active cycle of breathing techniques which includes cycle of breathing control, thoracic expansion exercises and forced expiratory technique (FET), appears to have beneficial effects.

Rehabilitation exercise can lessen the possibility of the progressive exacerbation of the patient's condition, exerting an active role in improving their lung function and the quality of the patients' life. Therefore, researcher have designed a lung function exercise bottle, which is capable of adjusting the pressure according to the patient's needs. The blowpipe can be inserted into the bottle body and the patient can blow the air through the tube. the air pressure in the bottle can be adjusted, with the advantage of wider range of application, lower cost and more convenient.

Secretion production and retention is top most complication of chronic obstructive pulmonary disease. First step of its management is removal of secretion as soon as possible to prevent infection and development of further complications. ACBT is one of most commonly used technique used in all times. But blow bottle is not only economic but also provide direct visual stimulus during performance to enhance patient interest. So it is necessity to find out the comparison of these two technique which will help to get the better quality of life, reduce the severity of disease and improve the pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Moderate COPD
* Hx of chronic sputum production
* Regular expectoration
* After 48 hours of admission in hospital
* Patient of 45 to 65 years
* Both genders (male and female)

Exclusion Criteria:

* Pulmonary disease like, Bronchiectasis, pneumothorax, TB, atelectasis
* Lung Abscess
* Lung cancer
* Any post-surgical (pneumectomy, lobectomy)
* Hemoptysis

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Breathlessness, Cough and Sputum Scale (BCSS). | 5thy day
  This scale is used to measure severity of breathlessness, cough and sputum. It is consist of 5 levels 0 to 4. In which 0 means unaware of difficulty,1 means mild,2 means moderate, 3 means marked and 4 means severe difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Zia, phd*, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petty TL. The history of COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(1):3-14. doi: 10.2147/copd.2006.1.1.3. PMID 18046898
- [Background] Gerayeli FV, Milne S, Cheung C, Li X, Yang CWT, Tam A, Choi LH, Bae A, Sin DD. COPD and the risk of poor outcomes in COVID-19: A systematic review and meta-analysis. EClinicalMedicine. 2021 Mar;33:100789. doi: 10.1016/j.eclinm.2021.100789. Epub 2021 Mar 18. PMID 33758801
- [Background] Brashier BB, Kodgule R. Risk factors and pathophysiology of chronic obstructive pulmonary disease (COPD). J Assoc Physicians India. 2012 Feb;60 Suppl:17-21. No abstract available. PMID 23155808
- [Background] Adeloye D, Song P, Zhu Y, Campbell H, Sheikh A, Rudan I; NIHR RESPIRE Global Respiratory Health Unit. Global, regional, and national prevalence of, and risk factors for, chronic obstructive pulmonary disease (COPD) in 2019: a systematic review and modelling analysis. Lancet Respir Med. 2022 May;10(5):447-458. doi: 10.1016/S2213-2600(21)00511-7. Epub 2022 Mar 10. PMID 35279265
- [Background] Kamal R, Srivastava AK, Kesavachandran CN, Bihari V, Singh A. Chronic obstructive pulmonary disease (COPD) in women due to indoor biomass burning: a meta analysis. Int J Environ Health Res. 2022 Jun;32(6):1403-1417. doi: 10.1080/09603123.2021.1887460. Epub 2021 Feb 12. PMID 33573386
- [Background] Rajnoveanu AG, Rajnoveanu RM, Motoc NS, Postolache P, Gusetu G, Man MA. COPD in Firefighters: A Specific Event-Related Condition Rather than a Common Occupational Respiratory Disorder. Medicina (Kaunas). 2022 Feb 5;58(2):239. doi: 10.3390/medicina58020239. PMID 35208563
- [Background] Halbert RJ, Isonaka S, George D, Iqbal A. Interpreting COPD prevalence estimates: what is the true burden of disease? Chest. 2003 May;123(5):1684-92. doi: 10.1378/chest.123.5.1684. PMID 12740290
- [Background] Medrinal C, Bonnevie T. [Physiotherapy during and after acute exacerbation of COPD]. Rev Mal Respir. 2022 Apr;39(4):386-397. doi: 10.1016/j.rmr.2022.02.056. Epub 2022 Feb 24. French. PMID 35221161
- [Background] Mansha H, Rashid S, Khalid MU, Khan RR, Hassan M, Khalid H. Effects of Active Cycle of Breathing Techniques on quality of life in patients with Chronic Bronchitis. Foundation University Journal of Rehabilitation Sciences. 2022;2(2):40-5.
- [Background] Liu H, Zhang X, Zhang Y. [Design and application of a pulmonary function exercise bottle]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2019 Feb;31(2):236-237. doi: 10.3760/cma.j.issn.2095-4352.2019.02.023. Chinese. PMID 30827317
- [Background] Zisi D, Chryssanthopoulos C, Nanas S, Philippou A. The effectiveness of the active cycle of breathing technique in patients with chronic respiratory diseases: A systematic review. Heart Lung. 2022 May-Jun;53:89-98. doi: 10.1016/j.hrtlng.2022.02.006. Epub 2022 Feb 27. PMID 35235877
- [Background] Hichkad S, Ganesh B. Effect of blow bottle device and flutter on functional capacity, dyspnea, fatigue, and peak expiratory flow rate in mild-to-moderate COPD patients: A comparative study. Indian Journal of Respiratory Care. 2021;10(3):294.
- [Background] Pakpahan R, Tarigan AP. The Effect of the Combination of Chest Physiotherapy and Active Cycle Breathing Technique on Respiratory Rate and Ability to Expend Sputum in Chronic Exacerbation Obstructive Lung Disease Patients at Haji Adam Malik Hospital Medan. European Journal of Molecular & Clinical Medicine. 2021;8(3):616-23.
- [Background] Zuriati Z, Surya M. Effectiveness Active Cycle of Breathing Technique (ACBT) with Pursed Lips Breathing Technique (PLBT) to tripod position in increase oxygen saturation in patients with COPD, West Sumatera. Enfermeria Clinica. 2020;30:164-7.
- [Background] Shen M, Li Y, Ding X, Xu L, Li F, Lin H. Effect of active cycle of breathing techniques in patients with chronic obstructive pulmonary disease: a systematic review of intervention. Eur J Phys Rehabil Med. 2020 Oct;56(5):625-632. doi: 10.23736/S1973-9087.20.06144-4. Epub 2020 May 13. PMID 32397703
- [Background] Gulati M, Singh K, Yadav H, Kumar S, Verma A. An Immediate Effect of Conventional Physiotherapy versus ACBT with Autogenic Drainage on Dyspnoea and Cough in Patient with COPD-A Randomized Control Trial.
- [Background] Katke S, Anthikat M. Comparative Study of Flutter Device and Active Cycle of Breathing Technique in Airway Clearance in Subjects with Chronic Obstructive Pulmonary Disease. Website: www ijpot com. 2020;14(3):232.